CLINICAL TRIAL: NCT06253910
Title: Comparison of Free Gingival Graft and Modified Apical Repositioning Flap Techniques to Create Attached Gingiva: A Long-Term (2 Year) Retrospective Study
Brief Title: Comparison of Free Gingival Graft and Modified Apical Repositioning Flap Techniques
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: waiting for re-calls
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Nur Balci, DDs, PhD, Associate Prof Dr, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 79
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Periodontal Diseases
Keywords: attached gingiva; free gingival graft
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patient selection (Other): A total of 15 (female) patients, between 31 and 70 years, who were systemically and periodontally healthy and applied to the periodontology clinic for treatment, were included in our study. Criteria for inclusion in the study are having ≥15 permanent teeth excluding third molars, not using any orthodontic appliance, not being pregnant or breastfeeding, not having any uncontrolled chronic and/or auto-immune disease, and not smoking.
  Interventions: Other: Patients selection
- MARF and FGG tehcniques (Other): Free gingival graft for the treatment of a total of 21 teeth with gingival recession in the lower jaw incisors area, no bone dehiscence, and the amount of attached gingiva being at least 0.5 mm and at most 1.5 mm and modified apically positioned flap methods were randomly selected (coin toss) and applied by a single investigator (MY). Surgical methods were performed on a minimum of 1 and a maximum of 2 teeth in the treated areas.
  Interventions: Other: Patients selection
- Post-surgical evalution and periodontal measurements (Other): Clinical periodontal parameters (plaque index (PI), pocket probing depth (PPD), bleeding on probing (BOP), gingival recession (GR) and clinical attachment level (CAL)) were recorded and evaluated at baseline, third months, first and second years. Periodontal measurements (keratinized tissue width (KTW), attached gingiva width (AGW)) recorded and evaluated at baseline, third months, first and second years.
  Interventions: Other: Recall visits

INTERVENTIONS:
Other: Patients selection — Patient selection were selected according to selected criteria.
  Arms: MARF and FGG tehcniques; Patient selection
Other: Recall visits — Following the operations, periodontal measurements were measured at the baseline, third month, first and second years.
  Arms: Post-surgical evalution and periodontal measurements

SUMMARY:
Attached gingiva, a crucial component of the keratinized tissue, plays a vital role in preserving periodontal health. The free gingival graft (FGG) and modified apically repositioned flap (MARF) techniques are frequently used for addressing issues related to insufficient attached gingiva. The aim of this study was to compare the efficiency of the FGG and the MARF increasing the zone of attached gingiva in 2-year posttreatment.

DETAILED DESCRIPTION:
The study included 15 participants who were both systemically and periodontally healthy, and these participants had a total of 21 teeth (10 for SDG and 11 for MARF). All included teeth had an attached gingiva width ranging from 0.5 mm to 1.5 mm and showed no signs of bone dehiscence. SDG and MARF methods were selected randomly (coin-to-coin). Clinical parameters recorded at baseline, third month, at first and second years were plaque index (PI), pocket probing depth (PPD), keratinized tissue width (KTW), attached gingiva width (AGW), bleeding on probing (BOP), gingival recession (GR) and clinical attachment level (CAL).

ELIGIBILITY:
Inclusion Criteria:

* having ≥15 permanent teeth excluding third molars,
* not using any orthodontic appliance,
* not being pregnant or breastfeeding,
* not having any uncontrolled chronic and/or auto-immune disease,
* not smoking.

Exclusion Criteria:

* having chronic and/or auto-immune disease
* smoking.

Ages: 34 Years to 58 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Attached gingiva width | Baseline, third month, first year and second years.
  The width of the attached gingiva was calculated by measuring the distance from the crest of the gingival margin to the mucogingival junction and then subtracting the probing depth of the gingival sulcus from this distance on the particular tooth.
Keratinized tissue width | Baseline, third month, first year and second years.
  The width of the keratinized tissue was calculated by measuring the distance from the crest of the gingival margin to the mucogingival junction

SECONDARY OUTCOMES:
Pocket probing depth | Baseline, third month, first year and second years.
  Measurement of the depth of a sulcus or periodontal pocket determined by measuring distance from a gingival margin to the base of the sulcus or pocket with a calibrated periodontal probe.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, School of Dentistry, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- [Background] Carnio J, Camargo PM, Klokkevold PR, Pirih FQ. The Modified Apically Repositioned Flap Technique: A Long-Term (4 to 16 Years) Retrospective Study. Int J Periodontics Restorative Dent. 2018 July/August;38(4):519-524. doi: 10.11607/prd.3028. Epub 2017 Dec 15. PMID 29244886
- [Background] Carnio J, Carnio AT, Pirih FQ, Cordero MG, Camargo PM. The Modified Apically Repositioned Flap Technique and Its Potential to Create Attached Gingiva in Areas with No Keratinized Tissue: A Long-Term (1 to 11 Years) Retrospective Case Series Study. Int J Periodontics Restorative Dent. 2020 Jan/Feb;40(1):103-109. doi: 10.11607/prd.4241. PMID 31815979
- See also: for discussion — https://pubmed.ncbi.nlm.nih.gov/22669155/
- See also: for discussion — https://pubmed.ncbi.nlm.nih.gov/29244886/